CLINICAL TRIAL: NCT01091168
Title: Phase III Trial of IV Vinflunine Versus an Alkylating Agent in Patients With Metastatic Breast Cancer Previously Treated With or Resistant to an Anthracycline, a Taxane, an Antimetabolite, and a Vinca-alkaloid (Study L00070 IN 308 B0)
Brief Title: Trial of Vinflunine Versus Alkylating Agent in Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L00070 IN 308 B0
Record Dates: First submitted 2010-02-03; First posted 2010-03-23 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm A: Vinflunine (Experimental): Patients randomised in the test arm (arm A) received VFL at the dose of 280 mg/m² on day 1 of each cycle every 3 weeks, over a 20-minute intravenous (IV) infusion. Cycles were repeated every 3 weeks.
  Interventions: Drug: vinflunine
- arm B: Alkylating agent of physician choice (Active Comparator): Patients randomised in the control arm (arm B) received an alkylating agent used as a single agent which was available in the investigational center and was approved for the treatment of cancer in the country.
  Interventions: Drug: Alkylating agent of physician choice registered in cancer

INTERVENTIONS:
Drug: vinflunine — 280 mg/m2 on day 1 of each cycle every 3 weeks
  Other Names: JAVLOR; L00070
  Arms: arm A: Vinflunine
Drug: Alkylating agent of physician choice registered in cancer — cyclophosphamide or melphalan or mitomycin C or thiotepa or cisplatin or carboplatin
  Other Names: Various
  Arms: arm B: Alkylating agent of physician choice

SUMMARY:
In metastatic breast cancer (MBC) patients who have already received anthracyclines, taxanes, antimetabolites and vinca-alkaloids and have developed drug resistance to these drugs, therapeutic options are very limited. Alkylating agents showed a modest activity in pretreated metastatic breast cancer. This phase III trial will compare the effectiveness and the safety profile of vinflunine to an alkylating agent of physician choice in MBC patients who have exhausted anthracyclines, taxanes, antimetabolites and vinca-alkaloids.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer in women worldwide and the second leading cause of cancer-related deaths in women.

Patients with metastatic breast cancer (MBC) remains incurable, and current goals of therapy are to ameliorate symptoms, delay disease progression, improve or at least maintain quality of life (QoL), and prolong overall survival (OS).There are a number of agents with established single-agent activity, with the anthracyclines and taxanes considered generally the most active. In addition, several drugs with different mechanisms of action such as antimetabolites and vinca-alkaloids have also demonstrated substantial activity in the metastatic setting as single-agents or in combination.

In patients who progress after having received anthracyclines, taxanes, antimetabolites and vinca- alkaloids, therapeutic options are scarce. In this heavily pretreated population for whom overall survival is not expected to exceed 6 to 7 months, there is a clear need for novel therapies.

Vinflunine (VFL) is a microtubule inhibitor obtained by semi-synthesis, interacts with tubulin at the vinca-binding domain and inhibits tubulin assembly by perturbing microtubule dynamics and mitotic spindles without affecting assembled microtubules. VFL antitumour activity was fully demonstrated against a large and varied panel of murine and xenograft models.

The main haematological toxicity reported was the neutropenia Grade 3-4 (40-50%). The incidence of its complications (febrile neutropenia and neutropenic infection) was less than 8%. The main non-haematological toxicity Grade 3-4 (with an incidence more than 10%) reported were constipation and fatigue.

This was a prospective multicentre, open-label, randomised (1:1), phase III study comparing OS in patients treated with vinflunine versus those treated with an alkylating agent of physician's choice as third line treatment or more for patients with locally recurrent and/or metastatic breast cancer previously treated with and no longer candidate to anthracyclines, antimetabolites, taxanes and vinca- alkaloids..

The primary endpoint for the trial was OS. Patients were assessed for toxicity, tumour response and progression and status (alive-dead) at regular intervals during the study treatment and the follow-up period. Patients were treated until disease progression, unacceptable toxicity, patient or investigator's decision. After the study treatment discontinuation, patients were followed until death.

The VFL dose of 280 mg/m² was the selected dose for this phase III study in patients with heavily pre- treated MBC. Indeed, VFL dose was reduced from 320 to 280 mg/m² in advanced transitional cell carcinoma of urothelial tract patients with performance status (PS) of 1 or with PS of 0 and having received prior pelvic irradiation. This dose was more regularly tolerable in patients with advanced disease stage who were heavily pre-treated.

ELIGIBILITY:
Inclusion Criteria:(main conditions)

* Female patients 18 to 75 years of age with metastatic breast cancer histologically/cytologically confirmed not amenable to curative surgery or radiotherapy and who have received at least two prior chemotherapy regimens including anthracyclines,taxanes,antimetabolite and vinca-alkaloid and are no longer candidate for these drugs,
* Karnofsky performance score of at least 70 %, adequate haematological, hepatic and renal functions and ECG without clinically relevant abnormality.

Exclusion Criteria:

* Concurrent serious uncontrolled medical disorder,
* known or clinical evidence of brain metastases or leptomeningeal involvement,
* pulmonary lymphangitis or symptomatic pleural effusion or symptomatic ascites,
* history of second primary malignancy,
* HIV infection, preexisting neuropathy,
* pregnancy or breast feeding.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-08-27 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Keddad, MD, PhD, Study Director — Institut de Recherche Pierre Fabre
Locations (80):
- Argentina (5):
  - Buenos Aires
  - Quilmes
  - Rosario
  - San Martín
  - San Miguel de Tucumán
- Austria (3):
  - Graz
  - Salzburg
  - Vienna
- Belarus (4):
  - Grodno
  - Homyel
  - Minsk
  - Vitebsk
- Belgium (3):
  - Brussels
  - Haine-Saint-Paul
  - Yvoir
- France (20):
  - Angers
  - Brest
  - Clermont-Ferrand
  - Dijon
  - Grenoble
  - Le Mans
  - Lille
  - Limoges
  - Lorient
  - Montpellier
  - Nancy
  - Nantes
  - Nice
  - Paris
  - Pontoise
  - Reims
  - Rouen
  - Saint-Brieuc
  - Saint-Priest-en-Jarez
  - Strasbourg
- Germany (6):
  - Berlin
  - Dortmund
  - Essen
  - Mainz
  - Munich
  - Trier
- Italy (7):
  - Ancona
  - Aviano
  - Bolzano
  - Brindisi
  - Frattamaggiore
  - Macerata
  - Orbassano
- Lisbon, Portugal
- Russia (10):
  - Arkhangelsk
  - Engel's
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Stavropol
  - Tambov
  - Ufa
  - Volgograd
- South Africa (3):
  - Durban
  - Johannesburg
  - Pretoria
- Spain (4):
  - A Coruña
  - Barcelona
  - Madrid
  - Seville
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan District
- Ukraine (4):
  - Dnipropetrovsk
  - Kharkiv
  - Khmelnytskyi
  - Kyiv
- United Kingdom (7):
  - Burnley
  - Cornwell
  - Derby
  - Glasgow
  - Ipswich
  - Preston
  - Worthing

REFERENCES:
- [Derived] Cortes J, Perez-Garcia J, Levy C, Gomez Pardo P, Bourgeois H, Spazzapan S, Martinez-Janez N, Chao TC, Espie M, Nabholtz JM, Gonzalez Farre X, Beliakouski V, Roman Garcia J, Holgado E, Campone M. Open-label randomised phase III trial of vinflunine versus an alkylating agent in patients with heavily pretreated metastatic breast cancer. Ann Oncol. 2018 Apr 1;29(4):881-887. doi: 10.1093/annonc/mdy051. PMID 29481630

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinflunine (VFL): Patients randomised in the test arm (arm A) received Vinflunine at the dose of 280 mg/m² on day 1 of each cycle every 3 weeks, over a 20-minute intravenous (IV) infusion. Cycles were repeated every 3 weeks.
  vinflunine: 280 mg/m2 on day 1 of each cycle every 3 weeks
- Alkylating Agent: Patients randomised in the control arm (arm B) received an alkylating agent used as a single agent which was available in the investigational center and was approved for the treatment of cancer in the country.
  Alkylating agent of physician choice registered in cancer: cyclophosphamide or melphalan or mitomycin C or thiotepa or cisplatin or carboplatin
Period: Overall Study
Arm/Group | Vinflunine (VFL) | Alkylating Agent
Started | 298 | 296
Completed | 0 | 0
Not Completed | 298 | 296
Not completed — Progressive disease | 250 | 234
Not completed — Adverse Event | 21 | 24
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician, patient's decision, other | 27 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Vinflunine | Arm B: Alkylating Agent of Physician Choice | Total
Number analyzed (Participants) | 298 | 296 | 594
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 236 | 227 | 463
  >=65 years | 62 | 69 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 296 | 594
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The main endpoint of this study is overall survival defined as the time from randomisation to the date of death or last follow-up. For patients who have not died, survival duration will be censored at the date of last contact or last follow-up or the date of last news.
Time Frame: From baseline up to 3 years 1 month
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Vinflunine: Patients randomised in the test arm (arm A) received VFL at the dose of 280 mg/m² on day 1 of each cycle every 3 weeks, over a 20-minute intravenous (IV) infusion. Cycles were repeated every 3 weeks.
  vinflunine: 280 mg/m2 on day 1 of each cycle every 3 weeks
Arm/Group | Vinflunine | Alkylating Agent
Number analyzed (Participants) | 298 | 296
Months | 9.1 [7.7 to 10.4] | 9.3 [7.5 to 10.9]
Statistical Analysis 1: Comparison: Vinflunine vs Alkylating Agent; Kaplan-Meier curves and life tables by treatment arm were provided. Confidence intervals on the median were calculated using the Brookmeyer and Crowley method. Hazard ratio and 95% confidence intervals were reported. A stratified Cox proportional model was performed to compare the two treatment arms taking into account the stratification factors (except centre) used at the time of randomisation; Test type: Superiority; p = 0.673, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.86 to 1.25]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of patients with Complete Response (CR), Partial Response (PR) and stable disease (SD), relative to the total number of patients in the analysed population.
Time Frame: From baseline up to 3 years 1 month
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vinflunine | Alkylating Agent
Number analyzed (Participants) | 298 | 296
Percentage of participants | 43.6 [37.9 to 49.3] | 35.5 [30 to 41.2]
Statistical Analysis 1: Comparison: Vinflunine vs Alkylating Agent; The disease control rate (DCR) were compared in the ITT population and in the population evaluable for response between the 2 arms with a cochran Mantel Haenszel, stratified on WHO performance status at baseline, number of prior chemotherapy lines for the treatment of disease and disease measurability at Baseline; Test type: Superiority; p = 0.0424, Log Rank

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomisation to the first tumour progression or death due to any cause in the absence of previous documentation of objective tumour progression. PFS was performed in the ITT and eligible populations every 6 weeks based on RECIST version 1.1. For patients lost of follow up, or without a known record of progression or death, PFS was censored at the date of last tumour assessment or the date of last contact of a follow-up showing no progression which ever occured last.
Time Frame: From baseline to cut-off date(27 August 2012), up to 3 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine | Alkylating Agent
Number analyzed (Participants) | 298 | 296
Months | 2.5 [1.7 to 2.7] | 1.9 [1.5 to 2.6]
Statistical Analysis 1: Comparison: Vinflunine vs Alkylating Agent; PFS was compared between the 2 treatment arms by the log-rank test procedure with the 5 % significant level, stratified on the stratification factors (except study site) as specified at the time of randomisation. Os was analysed using Kaplan-Meir method and summarized with median and 95% CI of the median; Test type: Superiority; p = 0.4927, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.8 to 1.12]

ADVERSE EVENTS:
Time Frame: Adverse events are reported from time of first dose of study treatment up to 30 days after last dose of study treatment (max treatment duration: 90 weeks) at the exception of Serious Adverse Events (SAE) occured after discontinuation and start of a further treatment, up to 4 years. AEs were collected from treated patients who received at least one study medication (N= 297 in vinflunine arm and N=290 in alkylating agent arm).
Description: The same event may appear as both an AE and SAE. However what is presented are distinct events. An event may be categorized as serious in 1 subject and as non serious in another. Specific AE tables were generated separately as per Eu format. we report here all "on study" SAEs and treatment related AEs by SOC and PT ( PT >=1%)
Arm/Group | Vinflunine | Alkylating Agent
All-Cause Mortality (participants affected / at risk) | 276/298 | 274/296
Serious Adverse Events (participants affected / at risk) | 82/297 | 66/290
Other Adverse Events (participants affected / at risk) | 197/297 | 262/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine (N=297) | Alkylating Agent (N=290)
Neutropenia (Blood and lymphatic system disorders) | 6 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Endocardititis staphylococcal (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Ileus (Gastrointestinal disorders) | 3 | 0
Ileus paralytic (Gastrointestinal disorders) | 3 | 0
Stomatis (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Oesophagial stenosis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Femur fracture (General disorders) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 | 43
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Neutropenic infections (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Catheter related infections (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine (N=297) | Alkylating Agent (N=290)
Neutropenia (Blood and lymphatic system disorders) | 37 | 31
Thrombocyotopenia (Blood and lymphatic system disorders) | 3 | 39
Constipation (Gastrointestinal disorders) | 102 | 23
Nausea (Gastrointestinal disorders) | 70 | 67
Abdominal pain (Gastrointestinal disorders) | 66 | 16
Stomatitis (Gastrointestinal disorders) | 52 | 18
Vomiting (Gastrointestinal disorders) | 34 | 33
Diarrhoea (Gastrointestinal disorders) | 16 | 19
Asthenia (General disorders) | 89 | 43
Injection site reaction (General disorders) | 29 | 2
Fatigue (General disorders) | 23 | 25
Weight decreased (Investigations) | 26 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 21 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 3
Anorexia (Metabolism and nutrition disorders) | 31 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No